CLINICAL TRIAL: NCT02174302
Title: Ì-SPIES, Comparison of Cystoscopy Images in Four Different SPIES Modalities
Status: Completed | Type: Observational
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-6
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Comparison of Images of the Same Area in the Bladder in Four Different SPIES Modalities on a Tablet Computer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of Images of the same area in the bladder in four different SPIES modalities on a tablet computer. Participants are asked to delineate the area on the image suspect for malignancy as precise as possible with a stylus on the tablet screen. Delineated area(s) is/are captured. Time to start the drawing and total time per image are captured. Hereafter, an judgement of Image quality is asked on a scale of 0 to 10, 0 being worst possible and 10 being best possible.

DETAILED DESCRIPTION:
Karl Storz Company has recently introduced the Storz Professional Image Enhancement System. To evaluate the interpretation of cystoscopy images in different SPIES modalities a tablet program was developed. Images of 20 bladder areas were captured in 4 different SPIES modalities; white light, Clara&Chroma, Spectra A and Spectra B. Of each bladder area, one extra image was added to the program, so that a total of 100 images were interpreted.

Every image is shown 45 seconds on the tablet screen. Participants are asked to delineate with a stylus on the tablet the precise area they suspect to be malignant and would resect or treat. After they are done they go to the next slide and the time is stopped.After each image, participants are asked to judge the quality of the image on a scale of zero to ten, with zero being the worst and ten the best.After this judgement, the next image for interpretation is presented.

ELIGIBILITY:
Inclusion Criteria:

* urologist or resident urologist

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: urologists and resident urologist
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Intra observer variability in delineated areas between the same bladder areas in different SPIES modalities. | 1 hour
Inter observer variability in delineated areas between the same bladder areas in different SPIES modalities. | 1 hour
Image quality of images in different SPIES modalities | 1 hour

SECONDARY OUTCOMES:
Differences in time to start delineation between images in different SPIES modalities | 1 hour
Differences in time needed per image in different SPIES modalities | 1 hour
Differences in use of úndo' button between different SPIES modalities | 1 hour
Differences in participants who are familiar with image enhancement system (NBI/SPIES) vs participants who are not familiar working with them. | 1 hour
Differences in interpretation of images between participants with a visual impairment or colourblindness vs participants without. | 1 hour
Differences in interpretations between participants in age or experience in TURBT annually. | 1 hour

REFERENCES:
- See also: Related Info — http://www.croesoffice.org